CLINICAL TRIAL: NCT00754793
Title: Sinusitis and Facial Pain Disorders Anti-Depression Trial
Acronym: SFPAT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Greg Davis, Assistant Professor, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 33501-B; 1KL2RR025015-01 (NIH); 1KL2RR025015-01 (NIH)
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Sinusitis; Facial Pain Disorder; Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): escitalopram 10mg - 30mg daily
  Interventions: Drug: escitalopram
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: escitalopram — 10mg - 30mg daily titrated as tolerated over 12 weeks
  Other Names: Lexapro (escitalopram)
  Arms: 1
Drug: placebo — inactive comparator; titrated as per protocol over 12 weeks
  Arms: 2

SUMMARY:
The study hypothesis is that the addition of an antidepressant to the standard treatment regimen in patients with both chronic sinusitis and depression or facial pain disorders and depression will decrease the report of chronic sinusitis or facial pain symptom severity.

This is a stratified, randomized, double-blind, placebo-controlled study using the drug escitalopram for the treatment of depression in patients experiencing depression and chronic sinusitis or depression and facial pain disorders.

It is a 12-week study. Subjects will have a screening visit and then be followed up by phone weekly for four weeks and bi-weekly for 8 weeks.

DETAILED DESCRIPTION:
All patients presenting to the University of Washington Medical Center Sinus Clinic are screened for depression with the PHQ-9 as a standard of care in their evaluation, as well as a physical examination, nasal endoscopy, and CT scan. Those patients who meet diagnostic criteria for CRS and for major depression will then be treated with three weeks of maximal medical therapy. Maximal medical therapy includes three weeks of a second-line antibiotic (such as Augmentin, azithromycin, or a fluoroquinolone), possible oral steroids based on the presence of inflammation or polyps in the sinuses, and nasal saline irrigations. They will then follow up with Dr. Davis in one month from their initial evaluation. Those who still do not have significantly improved symptoms (considered medical failures) will be approached and introduced to the study by Dr. Davis's medical assistant and then referred to the research assistant for further discussion and offered enrollment and consent if entry criteria are met. Note that if patients present for their initial consultation and have received maximal medical therapy from the referring clinician within the past two months, then they will be approached for possible entry into the study at that time.

Patients presenting with complaints of facial discomfort will also be included. These people often present with subjective sinusitis-like symptoms that are not objectively supported by CT scan or endoscopy. These patients are referred to the Neurology Clinic and will be asked to defer their appt. for the duration of the study.

Both patients and clinician will be blinded to the drug assignment. Subjects will be stratified according to facial pain or chronic sinusitis and then randomization will be done by restricted block randomization. A letter will be sent to each patient's primary care provider explaining this trial and that their patient may be taking an anti-depressant or a placebo.

During the trial, the dose of escitalopram will start at 10mg per day for seven days followed by 20mg per day for fourteen days, then will be maintained or titrated up based on our study's titration protocol.

At the conclusion of three months of active drug, the patient will be given the opportunity to continue the medication through their primary care provider. A two week supply of the active anti-depressant will be available to buffer this transition for patient's randomized to escitalopram.

Data Collection Phase 0: Recruitment All patients who meet criteria of CRS and depression or facial pain and depression will be monitored to determine how many patients were excluded and for what reasons. This is imperative for Specific Aim 1, to collect the data necessary to eventually calculate sample size and recruitment times for a future definitive trial.

Phase I: Patient Baseline Initial clinical, radiographic, and co-morbid characteristics will be identified using questionnaires and a short personal interview (by the study research assistant) as described below immediately following the initial one-month follow-up visit with Dr. Davis

Phase II: Patient Follow-up Subjects will be followed closely with weekly phone calls from the research assistant for the first four weeks of the trial. During these events, the PHQ-9 will be administered and questions will be asked regarding adverse events and side effects. After this, subjects will be telephoned bi-weekly for the duration of the trial asking the same questions. In addition, at one month and three months after the initiation of the research drug, during the telephone interview, subjects will be administered four questionnaires: the SNOT-20, SF-12, PHQ-9, and the SCL-20. Chronic sinusitis subjects and facial pain subjects will complete identical forms as there is common symptom crossover.

ELIGIBILITY:
Inclusion Criteria:

* meet diagnostic criteria for chronic sinusitis
* meet diagnostic criteria for facial pain disorder
* meet criteria for major depressive disorder on the PHQ-9
* 18 years of age or older
* established primary care provider
* able to read and speak English

Exclusion Criteria:

* unable to give informed consent of unable to complete self-administered questionnaires due to cognitive impairment, language barriers or severe medical condition
* terminal illness or significantly immunocompromized
* complications from chronic rhinosinusitis
* presence of sinus tumor
* isolated sphenoid disease
* immotile cilia syndrome
* currently on anti-depressant or mood stabilizer med.
* diagnosis of bipolar disorder, schizophrenic disorders, paranoid disorders, or psychotic disorders NOS
* significant suicide risk
* history of hospitalization for mental disorders including psychosis or depression
* history of drug abuse within prev. 6 months or dependency on any drug, including alcohol
* pregnant or breast feeding
* women of child-bearing potential not currently using an approved method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg E Davis, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited patients with chronic sinusitis and depression (PHQ9>=10) who were not already on an antidepressant.
Pre-assignment Details: No adverse events. No exclusions post enrollment.
Groups:
- Active Drug (Lexapro): escitalopram 10mg - 30mg daily
- Placebo: Placebo drug
Period: Overall Study
Arm/Group | Active Drug (Lexapro) | Placebo
Started | 1 | 2
Completed | 1 | 1
Not Completed | 0 | 1
Not completed — voluntary withdrawn from study | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Drug (Lexapro) | Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (45) | 50 (50) | 48 (48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Sino-Nasal Outcome Test-20 (SNOT-20)
Time Frame: baseline, 1 month, 3 months
Arm/Group | Active Drug (Lexapro) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Active Drug (Lexapro) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes